CLINICAL TRIAL: NCT03362099
Title: Efficacy of Genetic Markers in Choosing Pharmacological Treatment for Smoking Cessation With Bupropion and Varenicline and Its Implications for Combining Drugs: Randomized Control Study.
Brief Title: Efficacy of the Use of Genetic Markers in the Choice of the Pharmacological Treatment of Smoking (GENTSMOKING)
Acronym: GENTSMOKING
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Jaqueline Scholz, Principal Investigator, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 6013381600000068
Record Dates: First submitted 2017-11-16; First posted 2017-12-05 (Actual); Last update posted 2022-12-21 (Actual); Status verified 2022-12

CONDITIONS: Smoking Cessation; Genetic Predisposition
Keywords: varenicline; bupropion
MeSH Terms: conditions — Smoking Cessation; Genetic Predisposition to Disease | interventions — Varenicline; Bupropion

STUDY DESIGN:
Intervention Model Description: The Patients will be randomized in two arms. 200 will be treated in the pharmacogenetic arm and 200 in the varenicline arm ( control ).
Who Masked: Participant, Care Provider
Masking Description: The patients are blinded when they use varenicline. The care provider who makes clinical visits of the protocol do not have access to randomizing list, therefore they are blinded for the use of varenicline indicated, but not for bupropion use.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group Varenicline (No Intervention): Patients randomized to this group will collect polymorphisms at time zero and will receive varenicline for smoking cessation. The polymorphism result will only be known at the end of the protocol. Varenicline dosage 0,5 mg once a day for 3 days, after this 0,5 mg twice a day until seven day .At day eight 1 mg twice a day until complete week twelve.
- Group Genetic (Active Comparator): The patients randomized to this arm will collect polymorphisms and could receive varenicline or bupropion or both depending on genetic polymorphisms for each one these drugs.
  Bupropiona dosage 150 mg once a day seven days, after twice a day until complete week twelve. Varenicline dosage 0,5 mg once a day for 3 days, after this 0,5 mg twice a day until seven day .At day eight 1 mg twice a day until complete week twelve.
  Interventions: Drug: Varenicline Tartrate or bupropion

INTERVENTIONS:
Drug: Varenicline Tartrate or bupropion — the drug treatment will be chosen related to the polymorphism. If the polymorphism is favorable to varenicline the patient will receive varenicline, If it is favorable to bupropion the patient will receive bupropion, if not favorable to varenicline and bupropion the patient will receive bupropion + varenicline. If the patient has both favorable polymorphisms he will receive bupropion. Bupropiona dosage 150 mg once a day seven days, after twice a day until complete week twelve. Varenicline dosage 0,5 mg once a day for 3 days, after this 0,5 mg twice a day until seven day .At day eight 1 mg twice a day until complete week twelve.
  Other Names: Varenicline Tartrate and bupropion
  Arms: Group Genetic

SUMMARY:
Smoking is the leading cause of avoidable death in the world. Smoking is associated with the development of cardiovascular and respiratory diseases, as well as being considered a leading cause of cancer death. Data show that smokers have increased cardiovascular risk in relation to former smokers, even in comparison with individuals who have had a long and intense history tobacco use.

Considering this scenario, some drugs are used in tobacco cessation therapy. The first-line anti-smoking treatments approved by the Food and drug administration ( FDA ) are nicotinic reuptake therapy, bupropion ( norepinephrine and dopamine reuptake inhibitor) and varenicline ( partial agonist of nicotinic receptors composed of subunits alpha4Beta2 ). A metanalysis of 16 clinical studies indicated that smokers treated with bupropion had a higher abstinence rate compared to those receiving placebo - Odds ratio (OR ) - of 1,97 for treatment success.

Varenicline is more effective compared to others smoking cessation drugs approved by the FDA, with an OR of 2,27 ( IC 95% 2,02-2,55 ) compared to placebo. However, Varenicline is much more expensive than bupropion.

Significant advances in genetics have made the variability of the individual response to drugs, as far as efficacy as well as the rate of adverse effects, begin to be specifically investigated through pharmacogenetics studies.

DETAILED DESCRIPTION:
The patients will be invited to take part in the study collection genetic´s materials in order to determinate the frequency of CHRNA4 AND CYP2B6.

The polymorphisms in genes involved in the coding of metabolized drug enzymes, in the variability of carrier proteins or receptors are at the heart of these investigations. The gene CHRNA4 is an important gene for anti-smoking pharmacogenetics studies because they encode the alpha 4 beta 2 subunits of acetylcholine- nicotinic receptors ( which is important target for an action of varenicline ) and CYP2B6 major isoenzyme that metabolizes the bupropion. Rocha et al found the association of polymorphisms CHRNA4rs1044396 with success in smoking cessation in patients treated with varenicline and Tomaz et al found an association between CYP2B6rs2279343 and efficacy of bupropion.

Patients with the CC genotype, for the polymorphism CHRNA4rs1044396, had a lower success rate in treatment with varenicline( 29,5% ), compared to those with CT or TT genotypes (50,9% ) ( P =0,07 , n=167 ). The CT or TT genotypes were associated with a higher risk - Odds ratio ( OR ) - of success ( OR=1,67, IC 95%=1,10-2,53,P=0,02), in a multivariate model. Patients with the genotype AA, for the polymorphism CYP2B6rs2279343, obtained a higher success rate in treatment with bupropion ( 48,0% ), compared to patients with the AG or GG genotypes ( 35,5% ) (P=0,05,n=237). The AA genotype was associated with higher odds ratios for treatment success (OR=1,92,IC 95%=1,08-3,42,P=0,03) ,in a multivariate model.

It is suggested that these polymorphisms influence the pharmacological response and may be important for the design of an individualized pharmacotherapy.

ELIGIBILITY:
Inclusion Criteria:

* smoking who wants to quit smoking, stable clinic diseases, depression or anxiety disorder stable for more than 3 months

Exclusion Criteria:

* contra indication for varenicline and or bupropion
* unstable psychiatric disorders.
* In the treatment of neoplastic diseases.
* Limitation to attend the medical visits

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 361 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2022-04-15 (Actual); Study Completion 2022-04-15 (Actual)

PRIMARY OUTCOMES:
Bupropion favorable genetic marker | week 4 -
  Abstinence Rate confirmed througth carbon monoxide concentration in exhalated air in favorable bupropion smokers vs control arm with varenicline
Varenicline favorable genetic marker | week 4
  abstinence rate confirmed through carbon monoxide concentration in exhalated air in favorable varenicline genetic marker vs unfavorable varenicline genetic marker

SECONDARY OUTCOMES:
Abstinence rate at week 12 | At week 12
  Evaluation of add therapy for quitting smoking considering favorable and unfavaroble genetics markers

OTHER OUTCOMES:
Safety evaluation | week 0 until week 12
  Adverse events according to subjects self-reported

CONTACTS AND LOCATIONS:
Overall Officials: Jaqueline R Scholz, MD.Phd, Principal Investigator — Heart Institute - University of São Paulo - Braziil
Locations (1):
- Ambulatório de Tratamento Tabagismo - Incor HCFMUSP, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tomaz PR, Santos JR, Issa JS, Abe TO, Gaya PV, Krieger JE, Pereira AC, Santos PC. CYP2B6 rs2279343 polymorphism is associated with smoking cessation success in bupropion therapy. Eur J Clin Pharmacol. 2015 Sep;71(9):1067-73. doi: 10.1007/s00228-015-1896-x. Epub 2015 Jul 8. PMID 26153084
- [Background] Rocha Santos J, Tomaz PR, Issa JS, Abe TO, Krieger JE, Pereira AC, Santos PC. CHRNA4 rs1044396 is associated with smoking cessation in varenicline therapy. Front Genet. 2015 Feb 27;6:46. doi: 10.3389/fgene.2015.00046. eCollection 2015. PMID 25774163
- [Derived] Gaya PV, Fonseca GWP, Tanji LT, Abe TO, Alves MJNN, de Lima Santos PCJ, Consolim Colombo FM, Scholz JR. Smoking cessation decreases arterial blood pressure in hypertensive smokers: A subgroup analysis of the randomized controlled trial GENTSMOKING. Tob Induc Dis. 2024 May 16;22. doi: 10.18332/tid/186853. eCollection 2024. PMID 38756738
- [Derived] Gaya PV, Santos JR, Tomaz PRX, Abe TMO, Nassif M Jr, Galas LG, Bellini BB, Moraes IR, Santos PCL, Correa PCRP, Scholz JR. Efficacy of bupropion and varenicline genetic markers in choosing pharmacological treatment for smoking cessation, and implications for combining drugs: A randomized controlled trial - GENTSMOKING. Tob Induc Dis. 2024 Apr 16;22. doi: 10.18332/tid/186072. eCollection 2024. PMID 38628555
- See also: CYP2B6 rs2279343 polymorphism is associated with smoking cessation success in bupropion therapy — https://link.springer.com/article/10.1007/s00228-015-1896-x?no-access=true#citeas
- See also: CHRNA4 rs1044396 is associated with smoking cessation in varenicline therapy — https://www.frontiersin.org/articles/10.3389/fgene.2015.00046/full